CLINICAL TRIAL: NCT00382655
Title: Prehospital Screening to Prevent Injury and Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: The John A. Hartford Foundation (Other); University of Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10019
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: All Conditions
Keywords: Prevention; Emergency Medical Services; Emergency Medical Technicians
MeSH Terms: interventions — Educational Status; Referral and Consultation

INTERVENTIONS:
Procedure: Education and referral

SUMMARY:
The goal of this project is to prevent injuries and diseases among older adults through the development and evaluation of a novel emergency medical services (EMS)-based screening program to identify preventable injuries and diseases and refer the identified injuries and diseases for intervention.

To prevent injuries and diseases among older adults, this study specifically aims to:

1. Evaluate the feasibility of an EMS-based primary prevention program that screens older adults for need of the influenza and pneumococcal vaccine and for risk of falling during emergency medical responses in a rural setting;
2. Evaluate the outcome of the EMT-implemented screening and education program by performing a 14-day telephone follow-up on older adults cared for by EMTs.

At the conclusion of this award, we will determine if an EMT-implemented primary prevention program for older adults is feasible and benefits the community.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older;
* Request assistance from intervention group EMS agency
* Request assistance from control group EMS agency
* Request assistance between February 2003 and June 2005

Exclusion Criteria:

* Institutionalized
* Previous inclusion in study
* Unable to communicate in English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 700
Dates: Start 2003-02; Study Completion 2005-08

PRIMARY OUTCOMES:
Receipt of immunizations
Changes to home to prevent falls

SECONDARY OUTCOMES:
Discussion with physician regarding preventable diseases
Recollection of receiving educational materials

CONTACTS AND LOCATIONS:
Overall Officials: Manish N. Shah, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Department of Emergency Medicine, Rochester, New York, United States